CLINICAL TRIAL: NCT00003882
Title: Phase I Dose Finding Study of Anhydrovinblastine Administered as a 1-Hour Infusion Every 3 Weeks to Patients With Advanced Solid Tumors
Brief Title: Anhydrovinblastine in Treating Patients With Advanced Recurrent Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Nithya Ramnath, MD, Roswell Park Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067049; RPCI-DS-9844
Record Dates: First submitted 1999-11-01; First posted 2004-01-27 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: anhydrovinblastine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of anhydrovinblastine in treating patients who have advanced recurrent solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose and assess the toxicity of anhydrovinblastine in patients with advanced refractory solid tumors. II. Assess the safety, pharmacokinetics, and efficacy of this treatment regimen in this patient population.

OUTLINE: This is a dose escalation study. Patients receive anhydrovinblastine IV over 1 hour on day 1. Courses are repeated every 3 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity. The dose of anhydrovinblastine is escalated in cohorts of 1-6 patients until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose that at which no more than 2 of 6 patients experience dose limiting toxicity. Patients are followed at 1 month after treatment, and then monthly until death.

PROJECTED ACCRUAL: Approximately 30 patients will be accrued for this study within 8 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced solid tumor unresponsive to existing therapy and for which no curative therapy exists No hematologic malignancies

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 10 g/dL Hepatic: SGOT and SGPT no greater than 2.5 times upper limit of normal (ULN) Alkaline phosphatase no greater than 2.5 times ULN (except with bone metastases) PT and PTT no greater than ULN Bilirubin no greater than ULN Renal: Creatinine no greater than ULN OR Creatinine clearance at least 60 mL/min Cardiovascular: No congestive heart failure, angina pectoris (even if medically controlled), uncontrolled hypertension, arrhythmias, elevated CPK or recent EKG changes At least one year since myocardial infarction Neurologic: No history of neurologic or psychiatric disorders (e.g., dementia, seizures) No concurrent peripheral neuropathy greater than grade 1 Other: Not pregnant or nursing Fertile patients must use effective contraception No active infection No active pancreatitis Amylase no greater than the upper limit of normal No other serious systemic disease

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior biologic therapy and recovered No concurrent immunotherapy No concurrent colony stimulating factors (unless evidence of neutropenic infection) Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks for nitrosourea or mitomycin) Prior taxanes and vinca alkaloids allowed with recovery (excluding alopecia any grade and peripheral neuropathy no greater than grade 1) No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy and recovered At least 6 weeks since prior extensive radiotherapy to greater than 20% of bone marrow No concurrent radiotherapy Surgery: Not specified Other: No other concurrent experimental drugs At least 30 days since other investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 1999-03; Primary Completion 2000-04 (Actual); Study Completion 2000-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nithya Ramnath, MD, Study Chair — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Result] Schwartz GN, Bong D, Leichman CG, et al.: Phase I evaluation of anhydrovinblastine in patients with advanced malignancies. [Abstract] Proc Am Assoc Cancer Res 41: 3895a, 2000.